CLINICAL TRIAL: NCT03911388
Title: Phase 1 Trial of Engineered HSV G207 in Children With Recurrent or Refractory Cerebellar Brain Tumors
Brief Title: HSV G207 in Children With Recurrent or Refractory Cerebellar Brain Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cannonball Kids' Cancer Foundation (Other); Treovir, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0688; R01FD006368 (FDA); NCI-2021-00011 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Neoplasms, Brain; Glioblastoma Multiforme; Glioblastoma of Cerebellum; Neoplasms; Astrocytoma; Astrocytoma, Cerebellar; Neuroectodermal Tumors; Neuroectodermal Tumors, Primitive; Cerebellar PNET, Childhood; Cerebellar Neoplasms; Cerebellar Neoplasms, Primary; Cerebellar Neoplasm, Malignant; Cerebellar Neoplasm Malignant Primary; Neoplasm Metastases; Neoplasm Malignant; Neoplasms, Neuroepithelial; Neoplasms, Germ Cell and Embryonal; Neoplasms by Histologic Type; Neoplasms, Glandular and Epithelial; Neoplasms, Nerve Tissue; Central Nervous System Neoplasms, Primary; Central Nervous System Neoplasms, Malignant; Nervous System Neoplasms; Neoplasms by Site; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Medulloblastoma Recurrent; HSV; Virus; Pediatric Brain Tumor; Nervous System Cancer; Primitive Neuroectodermal Tumor (PNET) of Cerebellum
Keywords: Brain Tumor, Recurrent; Glioma; Glioblastoma Multiforme; Gliosarcoma; Medulloblastoma; Anaplastic Astrocytoma; Oligodendroglioma; Rhabdoid Tumor; Ependymoma; Germ Cell Tumor; Choroid Plexus Carcinoma; Cerebral Primitive Neuroectodermal Tumor; Giant Cell Glioblastoma; Atypical teratoid/rhabdoid tumor; Secondary Malignant Cerebellar Tumor; Embryonal Tumor; Neoplasms; Oncolytic Virus Therapy; Virotherapy, Oncolytic; Immunotherapy; Central Nervous System Agents; Antineoplastic Agents; Pediatric; Pediatrics; Oncolytic; Virus; HSV; Herpes Virus; G207; Oncolytic Herpes Virus
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Neoplasms; Astrocytoma; Neuroectodermal Tumors; Neuroectodermal Tumors, Primitive; Medulloblastoma; Cerebellar Neoplasms; Neoplasm Metastasis; Neoplasms, Neuroepithelial; Neoplasms, Germ Cell and Embryonal; Neoplasms by Histologic Type; Neoplasms, Glandular and Epithelial; Neoplasms, Nerve Tissue; Central Nervous System Neoplasms; Nervous System Neoplasms; Neoplasms by Site; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Virus Diseases; Glioma; Gliosarcoma; Oligodendroglioma; Rhabdoid Tumor; Ependymoma; Choroid Plexus Carcinoma

STUDY DESIGN:
Intervention Model Description: A traditional 3 + 3 design will be used with four patient cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HSV G207 (Experimental): Single dose of HSV-1 (G207) infused through catheters into region(s) of tumor. If G207 is safe in the first cohort of patients, subsequent patients will receive a single dose of G207 infused through catheters into region(s) of tumor followed by a 5 Gy dose of radiation to the tumor given with 24 hours of virus inoculation.
  Interventions: Biological: G207

INTERVENTIONS:
Biological: G207 — Single dose of G207 infused through catheters into region(s) of tumor. If G207 is safe in the first cohort of patients, subsequent patients will receive a single dose of G207 infused through catheters into region(s) of tumor followed by a 5 Gy dose of radiation to the tumor (which includes progressive leptomeningeal disease or any site of gross tumor progressing in the brain parenchyma) within 24 hours of virus inoculation.
  Other Names: HSV G207

SUMMARY:
This study is a clinical trial to determine the safety of inoculating G207 (an experimental virus therapy) into a recurrent or refractory cerebellar brain tumor. The safety of combining G207 with a single low dose of radiation, designed to enhance virus replication, tumor cell killing, and an anti-tumor immune response, will also be tested.

Funding Source- FDA OOPD

DETAILED DESCRIPTION:
Outcomes for children with recurrent or progressive cerebellar malignant brain tumors are very poor, and there are a lack of effective salvage therapies once a patient fails standard treatments. G207 is an oncolytic herpes simplex virus-1 (HSV) that has been successfully engineered to introduce mutations in the virus that enable it to selectively replicate in and kill cancer cells, but not normal cells. Replication of G207 in the tumor not only kills the infected tumor cells, but causes the tumor cell to act as a factory to produce new virus. These virus particles are released as the tumor cell dies, and can then proceed to infect other tumor cells in the vicinity, and continue the process of tumor kill. In addition to this direct oncolytic activity, the virus engenders an anti-tumor immune response; the virus is immunogenic and produces a debris field which exposes cancer cell antigens to immune cells which can target other cancer cells. Thus, the oncolytic effect of the virus and the immune response that the virus stimulates provide a "one-two punch" at attacking cancer cells. In preclinical studies, a single 5 Gy dose of radiation within 24 hours of virus inoculation to the tumor increased virus replication and tumor cell killing.

The safety of G207 has been demonstrated in 3 phase I clinical trials involving adults with supratentorial high-grade gliomas adults at the University of Alabama (UAB) and in an ongoing (closed to accrual) phase I clinical trial involving children with recurrent supratentorial brain tumors at Children's of Alabama. In the adult trials, high doses (up to 3 x 10^9 plaque-forming units) of virus were safely injected directly into the tumor or surrounding brain tissue without serious toxicities. Radiographic and neuropathologic evidence of anti-tumor responses have been seen. Preclinical laboratory studies have demonstrated that a variety of aggressive pediatric brain tumor types are sensitive to G207.

This study is a phase I, open-label, single institution clinical trial of G207 alone or combined with a single low dose of radiation in children and young adults, ages 3 to 21 years, with recurrent or progressive cerebellar brain tumors. The primary goal is to determine safety. The secondary aims are to obtain preliminary information on the effectiveness of and immune response to G207. A traditional 3 + 3 design will be used with four patient cohorts. The first cohort will receive G207 alone, and the next cohorts will receive G207 at one of three doses followed by a 5 Gy dose of radiation to active areas of tumor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 36 months and < 22 years
* Pathologically proven malignant cerebellar brain tumor (including medulloblastoma, glioblastoma multiforme, giant cell glioblastoma, anaplastic astrocytoma, primitive neuroectodermal tumor, ependymoma, atypical teratoid/rhabdoid tumor, germ cell tumor, or other high-grade malignant tumor) which is progressive or recurrent despite standard care including surgery, radiotherapy, and/or chemotherapy. A pathologically proven secondary malignant cerebellar tumor without curative treatment options is eligible.
* Lesion must be ≥ 1.0 cm ≤ 3.0 cm in diameter and surgically accessible as determined by MRI. Larger tumors may be surgically debulked and treated if ≤ 3.0 cm after debulking
* Patients must have fully recovered from acute treatment related toxicities of all prior chemotherapy, immunotherapy or radiotherapy prior to entering this study.
* Myelosuppressive chemotherapy: patients must have received their last dose at least 3 weeks prior (or at least 6 weeks if nitrosurea)
* Investigational/Biologic agents: patients must have recovered from any acute toxicities potentially related to the agent and received last dose ≥ 7 days prior to entering this study (this period must be extended beyond the time during which adverse events are known to occur for agents with known adverse events ≥ 7 days). For viral therapy, patients must have received viral therapy ≥ 3 months prior to study entry and have recovered from all acute toxicities potentially related to the agent.
* Monoclonal antibodies: The patient must have received last dose ≥ 21 days prior.
* Radiation: Patients must have received their last fraction of craniospinal radiation (>24 Gy) or total body irradiation ≥ 3 months prior to study entry. Patients must have received focal radiation to symptomatic metastatic sites or local palliative radiation ≥ 28 days prior to study entry.
* Autologous bone marrow transplant: Patients must be ≥ 3 months since transplant prior to study entry.
* Normal hematological, renal and liver function (absolute neutrophil count > 1000/mm3, platelets > 100,000/mm3, prothrombin time (PT) or partial thromboplastin time (PTT) < 1.3 x control, creatinine within normal institutional limits OR creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal, total bilirubin < 1.5 mg/dl, transaminases < 3 times above the upper limits of the institutional norm)
* Patients < 16 years, Modified Lansky performance score ≥ 60; patients ≥ 16 years, Karnofsky performance score ≥ 60
* Patient life expectancy must be at least 8 weeks
* Written informed consent in accordance with institutional and FDA guidelines must be obtained from patient or legal guardian

Exclusion Criteria:

* Any treatment outside the allowable guidelines outlined in section 5.1.
* Diffuse, widespread, abnormal tumor pattern involving 3 or more lobes of the brain
* Acute infection, granulocytopenia or medical condition precluding surgery
* Pregnant or lactating females
* Diagnosis of encephalitis or CNS infection < 3 months prior, or receiving ongoing treatment for encephalitis, CNS infection or multiple sclerosis
* Tumor involvement which would require ventricular or brainstem inoculation or would require access through a ventricle in order to deliver treatment
* Required steroid increase within 1 week prior to G207 inoculation or patients requiring >2 mg of dexamethasone daily
* Known HIV seropositivity
* Concurrent therapy with any drug active against HSV (acyclovir, valacyclovir, penciclovir, famciclovir, gancyclovir, foscarnet, cidofovir) or any immunosuppressive drug therapy (except dexamethasone or prednisone).
* Other current malignancy
* Concurrent anticancer or investigational drug

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability as Measured by Frequency of Grade 3 or Above Adverse Events | Baseline to 15 years
  All events with a Grade 3 or above toxicity (defined by the CTCAE v5.0) will be tabulated by event and by relationship to G207.

SECONDARY OUTCOMES:
Immunologic Response | Baseline to 24 months
  HSV-1 antibody titers will be checked by ELISA prior to the administration of G207 and at regular intervals after treatment.
Virologic Shedding | Baseline to 15 years
  HSV-1 antibody titers will be checked by ELISA prior to the administration of G207 and at regular intervals after treatment.
Progression Free Survival | Baseline to 24 months
  Time after G207 administration to clinical and radiographic disease progression will be evaluated.
Overall Survival | Baseline to 60 months
  The overall survival for each patient receiving G207 will be calculated
Change in Performance (Ability to Perform Normal Activities) | Baseline to 24 months
  A modified Lansky score (for children under 16 years of age) or Karnofsky score (for children 16 and older) will be recorded pre-treatment and measured serially at regular intervals after treatment. The score is a standard performance score that measures overall function of the child with a scale range from 0 (lowest, poorest performance score) to 100 (highest, best performance).
Quality of Life (optional) | Baseline to 24 months
  Quality of life will be measured with questionnaires taken at baseline (before administration of G207) and at specified times thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Friedman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Children's of Alabama, Birmingham, Alabama
  - St. Louis Children's Hospital, St Louis, Missouri
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03911388/ICF_000.pdf